CLINICAL TRIAL: NCT04864444
Title: Mass Drug Administration With Dihydroartemisinin-piperaquine and Primaquine to Reduce Malaria in a Moderate-low Transmission Setting in Senegal: A Cluster Randomized Controlled Trial
Brief Title: Mass Drug Administration of Dihydroartemisinin-piperaquine + Single Low-dose Primaquine to Accelerate Toward Elimination Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: L'université de Thiès (Other); Programme National de Lutte contre le Paludisme (PNLP), Senegal (Unknown); Population Services International (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); US President's Malaria Initiative (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-29886
Record Dates: First submitted 2021-04-22; First posted 2021-04-28 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Malaria,Falciparum; Malaria
Keywords: Antimalarials; Mass drug administration; Dihydroartemsinin; Piperaquine; Primaquine; Parasitic Diseases
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Parasitic Diseases | interventions — Primaquine

STUDY DESIGN:
Intervention Model Description: This is a two-arm cluster randomized controlled trial. A total of 60 villages will be randomized to receive the intervention (three rounds of MDA with DHA-PPQ + SLD-PQ) or control (standard malaria control measures, including SMC) at a ratio of 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MDA with DHA-PPQ + SLD-PQ (Experimental): Participants in intervention villages will be given three rounds of MDA with DHA-PPQ and SLD-PQ. Prior to the intervention, participants will have received piperonyl butoxide (PBO) treated LLINs and proactive community case management. Unlike control villages, MDA-randomized villages will not receive SMC.
  Interventions: Drug: Dihydroartemisinin-piperaquine; Drug: Primaquine
- Standard malaria control interventions (No Intervention): Participants in the control villages will receive standard malaria control interventions as implemented by the Senegal PNLP. This will include the distribution of PBO LLINs, proactive case management, and SMC.

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine — DHA-PPQ will be given over the course of three consecutive days using 160mg/20mg or 320mg/40mg of dihydroartemisinin/piperaquine tablets. DHA-PPQ will be administered via age-based dosing. All three doses will be directly observed and given orally with water and without food.
  Other Names: Duo-Cotecxin
  Arms: MDA with DHA-PPQ + SLD-PQ
Drug: Primaquine — Primaquine will be given once with the first dose of DHA-PPQ. Primaquine will be administered in an aqueous solution according to age-based dosing guidelines.
  Arms: MDA with DHA-PPQ + SLD-PQ

SUMMARY:
This community-based cluster randomized controlled trial aims to evaluate the effectiveness of time-limited, community-wide mass drug administration (MDA) with dihydroartemisinin-piperaquine (DHA-PPQ) and single low-dose primaquine (SLD-PQ) on Plasmodium falciparum transmission compared to standard-of-care seasonal malaria chemoprevention (SMC). The study will be conducted in a moderate-to-low malaria transmission setting of Senegal with optimized malaria control measures (e.g., proactive community case management and piperonyl butoxide pyrethroid long-lasting insecticidal nets (PBO LLINS)).

DETAILED DESCRIPTION:
Over the past two decades in Senegal, the scale-up of malaria control measures [e.g., access to prompt testing and case management, LLINs, and SMC] has led to a 78% reduction in malaria incidence. However, gains have not been uniform, with lower transmission areas in the north implementing pre-elimination activities and higher transmission areas in the south implementing control interventions (including SMC). The purpose of this study is determine whether MDA will be able to rapidly reduce malaria incidence in areas of moderate-to-low malaria transmission of southern Senegal (where control activities are ongoing) so that the program can reorient their malaria strategy to implement elimination interventions in these settings.

The study aims to deliver three rounds of community-wide MDA with DHA-PPQ + SLD-PQ. MDA drugs will be administered over the course of three days. All three doses of DHA-PPQ will be given via supervised DOT (as per administration of SMC by national malaria guidelines) through a door-to-door approach.

The research objectives are:

1. To evaluate the impact of three rounds of MDA with DHA-PPQ and SLD-PQ on village-level confirmed malaria case incidence, malaria prevalence, and on reaching a target malaria incidence of <5 cases per 1000 person-years compared to standard-of-care SMC when provided in the context of optimized control (proactive community case management + PBO LLINs).
2. To determine the cost, coverage, operational feasibility, and acceptability of three rounds of MDA with DHA-PPQ and SLD-PQ compared to standard-of-care SMC.
3. To determine the impact of three rounds of MDA with DHA-PPQ and SLD-PQ compared to standard-of-care SMC on parasite population dynamics and drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥3 months
* Willingness to comply with trial procedures and written informed consent to be obtained at the beginning of the study

Exclusion Criteria:

* Severe illness or self-reported chronic illness (e.g., HIV, tuberculosis, heart/liver/kidney disease, and severe malnutrition)
* Known hypersensitivity to study drug

Additional exclusion criteria for DHA-PPQ:

* First trimester pregnancy assessed by history and/or urine pregnancy testing
* Concurrent artemisinin-based combination therapy (ACT) use
* Taking drugs that influence cardiac function or prolong QTc interval

Additional exclusion criteria for PQ:

* Pregnancy (any trimester) or currently breastfeeding an infant <6 months of age assessed by history and/or urine pregnancy testing
* <2 years of age

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10715 (Actual)
Dates: Start 2021-06-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Difference in village-level confirmed incidence of malaria | one year post-MDA
  Village-level malaria incidence will be defined as the number of individuals diagnosed with malaria through proactive case detection and passive malaria surveillance at the health facility-level over the total village population measured during census.

SECONDARY OUTCOMES:
Difference in parasite prevalence by microscopy during high malaria transmission season | 3 months after last round of MDA
  Parasite prevalence will be assessed via microscopy from samples obtained during cross-sectional survey conducted at the end of the transmission season.
Difference in parasite prevalence by polymerase chain reaction (PCR) during high malaria transmission season | 3 months after last round of MDA
  Parasite prevalence will be assessed via polymerase chain reaction from samples obtained during cross-sectional survey conducted at the end of the transmission season.
Difference in serological markers of recent infection | 3 months after last round of MDA
  Difference in seroprevalence from samples obtained during cross-sectional survey conducted at the end of the transmission season.
Difference in the change in prevalence of drug resistance markers | Change from baseline to endline; 1 year period
  Prevalence of drug resistance markers (K13 and plasmepsin copy number) will be assessed from samples taken during the baseline and endline cross-sectional surveys.
Difference in the change in prevalence of parasite population dynamics | Change from baseline to endline; 1 year period
  Prevalence of parasite population dynamics (multiplicity of infection) will be assessed from samples taken during the baseline and endline cross-sectional surveys.

OTHER OUTCOMES:
Population coverage of MDA | Up to 18 weeks
  Coverage will be measured as the proportion of people who received MDA divided by the total number of persons in the population at each MDA round.
Difference in the cost-effectiveness of MDA versus SMC | Up to 24 months
  Costs of MDA and optimized control will be collected throughout the study period. The incremental cost-effectiveness ratio (ICER) will be used to compare MDA to SMC.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis Ndiaye, MD PhD, Principal Investigator — Université de Thiès; Michelle Hsiang, MD MSc, Principal Investigator — University of California, San Francisco; Doudou Séne, MD, Principal Investigator — Senegal Programme National de Lutte contre le Paludisme (PNLP); Katharine Sturm-Ramirez, PhD, Principal Investigator — US President's Malaria Initiative/CDC
Locations (1):
- Tambacounda Health District, Tambacounda, Senegal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ba EKC, Roh ME, Diallo A, Gadiaga T, Seck A, Thiam S, Fogelson A, Gaye S, Diallo I, Lo AC, Diouf E, Ba OG, Gueye AB, Wu X, Milligan P, Kibuka T, Hama M, Eckert E, Thwing J, Bennett A, Gosling R, Hwang J, Sene D, Ba F, Cisse B, Sturm-Ramirez K, Hsiang MS, Ndiaye JL. Effect of mass drug administration on malaria incidence in southeast Senegal during 2020-22: a two-arm, open-label, cluster-randomised controlled trial. Lancet Infect Dis. 2025 Jun;25(6):656-667. doi: 10.1016/S1473-3099(24)00741-2. Epub 2025 Jan 9. PMID 39799956
- [Derived] Ba Konko Cire EH, Roh ME, Diallo A, Gadiaga T, Seck A, Thiam S, Gaye S, Diallo I, Lo AC, Diouf E, Ba OG, Gueye AB, Fogelson A, Wu X, Milligan P, Kibuka T, Hama M, Eckert E, Thwing J, Bennett A, Gosling R, Hwang J, Sene D, Ba F, Cisse B, Sturm-Ramirez K, Hsiang MS, Ndiaye JL. Mass drug administration to reduce malaria incidence in a low-to-moderate endemic setting: short-term impact results from a cluster randomised controlled trial in Senegal. medRxiv [Preprint]. 2024 Jul 18:2024.07.17.24310593. doi: 10.1101/2024.07.17.24310593. PMID 39072042